CLINICAL TRIAL: NCT06246721
Title: The Attitude and Success Rate of Women with Pelvic Organ Prolapse on Self-management of Vaginal Pessary: a Multi-centered Prospective Study
Brief Title: Attitude and Success Rate of Women with Pelvic Organ Prolapse on Self-management of Vaginal Pessary
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, CHAN SYMPHOROSA SHING CHEE, Doctor, Chief of Service (O&G), Clinical Associate Professor (honorary), Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2023.603
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects Agree Self-management Group (Active Comparator): Women with pelvic organ prolapse requires ring pessary for treatment. Those who agree to join the study and agree to learn how to self-management of vaginal pessary.
  Interventions: Behavioral: Self-management of vaginal pessary
- Subjects Refuse Self-management Group (Placebo Comparator): Women with pelvic organ prolapse requires ring pessary for treatment. Those who agree to join the study and refuse to learn how to self-management of vaginal pessary.
  Interventions: Behavioral: Self-management of vaginal pessary

INTERVENTIONS:
Behavioral: Self-management of vaginal pessary — Self-management of vaginal pessary

SUMMARY:
This is a prospective cohort study aims at assessing patient's attitude towards self-management of vaginal pessary, and identifying factors that affect patient's level of acceptance towards self-management.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a common gynaecological condition worldwide with significant morbidity. Use of vaginal pessary has been recommended by multiple national authorities such as NICE and ACOG as an effective conservative management to all patients suffering from POP. However, the use of vaginal pessary can also associate with risks such as increased vaginal discharge, discomfort, bleeding and ulcers. The long term follow-up for changing pessary also exerts a significant economic cost in the healthcare system. Self-management of vaginal pessaries helps improved patient satisfaction and their quality of life with a much lower complication rates. Nevertheless, the attitudes and knowledge in women about pessary use is reported to be deficient and warrant further study.

This is a prospective cohort study aims at assessing patient's attitude towards self-management of vaginal pessary, and identifying factors that affect patient's level of acceptance towards self-management.

Patients who suffers from pelvic organ prolapse requiring the use of ring pessary as treatment will be invited to join the study, with exclusion criteria.

Should patient agree to join the study, they will fill in a self-administered questionnaire focusing on various reasons and factors that may influence patients' attitude on the use of vaginal pessaries and also Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ) at different time intervals to assess the symptoms, severity of symptoms and their impact on a woman's activities and well-being. Both PFDI and PFIQ are reliable, valid and condition-specific symptoms and QoL instruments for women with pelvic floor disorders, . Chinese validated versions are available. The epidemiological background information, any significant medical disease, especially previous treatment and surgery for pelvic organ prolapse would be gathered from the patient and medical records, if any. Patient will then be divided into two intervention arms by patient's own choice: self management arms and traditional hospital-based care arm, after counselling on the pros and cons of the above options with written counselling material. For patients who agree to learn self-management of vaginal pessary, per vaginal exam and staging of prolapse will be assessed and documented using Pelvic Organ Prolapse Quantification system (POP-Q) by gynaecologists. Pelvic floor muscles contraction and symptom of stress incontinence will be assessed and documented. PVC ring pessary will be inserted in the recruitment session. For those who has been stable on ring pessary without complication, a silicon ring pessary of their size will be suggested. Participants will need to bring their own purchased silicon ring pessary for the teaching session. For patient who has never tried ring pessary, a PVC ring pessary will be fitted first.

For patient who does not agree to try self-management, routine clinical care with hospital-based management will be provided as per department protocol with changing of PVC ring pessary and follow-ups appointments.

A teaching session will be arranged for a 1-to-1 20-minute self-management education by doctors or incontinence nurses to patient who agrees to learn self-management. Patient will be taught on self-insertion/removal of the silicon ring pessary, and silicon ring pessary care techniques. Returned demonstration from patient will be carried out to ensure patient's competence in self-management. Hotline will be given to patient in case of any difficulties in self-management of vaginal pessary.

For patients who experience difficulty in self-management either from hotline call-backs or during 6-month follow-up session, a second teaching session will be offered to reinforce the self-management techniques if the patient agrees to continue learning self-management.

Follow up will be arranged in 6 months to review patient's pelvic floor disorder symptoms, look for and document any pessary-related complications, and PFDI and PFIQ will be repeated for quality-of-life assessment. The frequency of self replacement will also be explored. If patient is well on self-management of ring pessary, a second 6-monthly follow up will be arranged and again to review patient's pelvic floor disorder symptoms, look for and document any pessary-related complications, and PFDI and PFIQ will be repeated for quality-of-life assessment. The frequency of self-replacement will also be explored. Patient's satisfaction will be explored using Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

Patient who suffers from pelvic organ prolapse requiring use of vaginal ring pessary as treatment

Exclusion Criteria:

1. Physically dependent in their daily living
2. Limited physical dexterity due to medical conditions, for example: Parkinsonism or stroke
3. Pregnancy
4. Cognitive deficit preventing informed consenting procedure and self management
5. Age lower than 18

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients willing to learn self-management of vaginal pessary | Baseline
  Questionnaire on attitude and knowledge will be asked. Descriptive analysis will be used to study the attitude of women on self-management of vaginal pessary. Prevalence of patients willing to learn self-management of vaginal pessary will be calculated.

SECONDARY OUTCOMES:
Successful rate in self-management of vaginal pessary | 6 months follow up and 12 months follow up
  Outcome of self-replacement will be recorded in datasheet. Descriptive analysis will be used to study the outcome of self-management of vaginal pessary, successful rate of self-management will be calculated.
Patient's satisfaction on self-management of vaginal pessary | 6 months follow up and 12 months follow up
  Question about patient's satisfaction on vaginal pessary and willing to continue self-management will be asked. Descriptive analysis will be used to study patient's satisfaction on self-management of vaginal pessary.
Basic demographics questions | Baseline, 6 months follow up and 12 months follow up
  Basic demographics will be collected in datasheet.
Quality of life validated questionnaire (PFDI/PFIQ short form) | Baseline, 6 months follow up and 12 months follow up
  Quality of life related to pelvic floor disorders will be measured by answering validated questionnaire (PFDI/PFIQ short form).

CONTACTS AND LOCATIONS:
Overall Officials: Shing Chee Symphorosa CHAN, Principal Investigator — O&G, PWH
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No